CLINICAL TRIAL: NCT05158985
Title: Comparative Study Between Different Duty Cycles of Ultrasound Diclofenac Phonophoresis in Management of Chronic Lateral Epicondylitis: Randomized Controlled Trial
Brief Title: Comparative Study Between Different Duty Cycles of Ultrasound Diclofenac Phonophoresis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, basma osama, Principal Investigator, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6786
Record Dates: First submitted 2021-11-18; First posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Undefined
MeSH Terms: interventions — Phonophoresis; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group A (Experimental): diclofenac sodium phonophoresis using continuous ultrasound with a frequency of 1MHz, an intensity of 1.5W/Cm2 for 4 minutes
  Interventions: Other: phonophoresis
- group B (Experimental): diclofenac sodium phonophoresis using pulsed US with 1:1 duty cycle with a frequency of 1MHz, an intensity of 1.5W/Cm2 for 4 minutes
  Interventions: Other: phonophoresis
- group C (Experimental): diclofenac sodium phonophoresis using pulsed US with 1:4 duty cycle with a frequency of 1MHz, an intensity of 1.5W/Cm2 for 10 minutes
  Interventions: Other: phonophoresis
- group D (Experimental): exercises only in form of (strengthening, stretching and occupational exercises).
  Interventions: Other: exercises

INTERVENTIONS:
Other: phonophoresis — treatment
  Arms: group A; group B; group C
Other: exercises — treatment
  Arms: group D

SUMMARY:
Lateral epicondylitis is a tendinopathy injury involving the extensor muscles of the forearm. These muscles originate on the lateral epicondylar region of the distal humerus. the insertion of the extensor carpi radialis brevis is involved in most cases. Transdermal administration of an anti-inflammatory drug to specific area is one of the methods that used to decrease inflammation and increase cell metabolism

DETAILED DESCRIPTION:
Lateral epicondylitis is a soft-tissue lesion of the tendinous origin of the wrist extensor muscles at their origin on the lateral humeral epicondyle. The extensor carpi radialis brevis is the area of most pathologic changes. It begins as a microtear of the tendinous origin of the wrist extensor muscles and results in degeneration and reactive granulation tissue formation. Activities involving prolonged or repeated gripping, wrist extension, forearm supination, and pronation cause eventual failure of the affected portion of the tendon. The mechanical failure of the tendon results in an ensuring tendinitis and symptoms of lateral epicondylitis. It is aggravated with movements of the wrist, by palpation of the lateral side of elbow, or by contraction of extensor muscles of the wrist.

There are different treatment methods for lateral epicondylitis. Initially, lateral epicondylitis has been treated with ice, rest, counterforce tennis brace and/or non-steroidal anti-inflammatory drugs. But when the condition is not responding to initial treatment physical therapy is initiated

ELIGIBILITY:
Inclusion Criteria:

1. Both sexes will be involved
2. Duration of the disease is more than 12 weeks.
3. Patient's age ranges from 20 to 40 years

Exclusion Criteria:

1. Diabetic patients.
2. Hypertension patients.
3. Pregnant women
4. Cardiovascular patients
5. Patients with malunion fractures
6. Patients with cervical Radiclopathy
7. Patients with olecranon bursitis

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2020-05-15 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale for pain intensity measurement | 4 weeks
  A VAS is usually a horizontal line, 100 mm in length, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain". The patient marks on the line the point that they feel represents their perception of their current state
Hand grip dynamometer for hand grip measurement | 4 weeks
  The dynamometer has a dual scale readout which displays isometric grip force from 0-90 kg (0-200 lb). The outer dial registers the result in kg and the inner dial registers the result in lb. It has a peak hold needle which automatically retains the highest reading until the device is reset. The handle easily adjusts to five grip positions from 35-87 mm (1½ - 3¼") in 13 mm (½") increments. Always use the wrist strap to prevent the dynamometer from falling on the floor if accidentally dropped

CONTACTS AND LOCATIONS:
Locations (1):
- Emad MOHAMED, Cairo, Egypt